CLINICAL TRIAL: NCT01077011
Title: Acute Comfort and Blur Profile of a Lubricant Eye Drop Versus a Marketed Lubricant Eye Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C-09-060
Record Dates: First submitted 2010-02-18; First posted 2010-02-26 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubricant eye drop (Experimental): Lubricant eye drop
  Interventions: Other: Lubricant eye drop FID 115958D
- GenTeal Gel (Active Comparator): GenTeal Gel
  Interventions: Other: GenTeal Gel

INTERVENTIONS:
Other: Lubricant eye drop FID 115958D — 1 drop in each eye, one time
  Arms: Lubricant eye drop
Other: GenTeal Gel — 1 drop in each eye, one time
  Arms: GenTeal Gel

SUMMARY:
The purpose of this study is to compare the comfort and blurriness of an investigational lubricant eye drop with a marketed lubricant eye gel.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye

Exclusion Criteria:

* Must not have worn contact lenses within 12 hours preceding enrollment
* Must not have used any topical ocular drops or ointment within 24 hours preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Three-minute visual blur profile | Through 3 minutes (post-instillation)
Overall Acceptability | Immediately upon instillation

SECONDARY OUTCOMES:
Drop Comfort Upon Instillation | Immediately upon installation

REFERENCES:
- [Result] http://www.aaopt.org/evaluation-efficacy-and-patient-acceptance-new-lubricant-eye-gel